CLINICAL TRIAL: NCT05949372
Title: The Effect of Two Different Breastfeeding Positions on Breastfeeding Self-efficacy, Breastfeeding Success and Postpartum Comfort in Primiparous Mothers.
Brief Title: The Effect of Breastfeeding Position on Breastfeeding Self-efficacy, Success and Postpartum Comfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, dilek menekşe, Assistant professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sema Aktaş
Record Dates: First submitted 2023-06-28; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Breastfeeding
Keywords: Breastfeeding position; football hold; biological breastfeeding; biological nuturing
MeSH Terms: conditions — Breast Feeding | interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single-blind (researchers are not blinded) randomization will be provided, as the breastfeeding position will be given to the mother and newborn by the researchers. The statistician was also blinded for the data analysis purpose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group : (Biological Breastfeeding Position) (Experimental): The first breastfeeding after birth will take place within the first half hour - two hours. The second breastfeeding will be performed 2 hours after the first breastfeeding, and the third breastfeeding will be performed at the 24th hour. Three measurements will be made in total.The mother is half-sitting, in the most comfortable position where she can make eye contact with her baby. The baby's head is placed on the mother's chest with her legs on the mother's stomach. With this position, gravity fixes the baby's whole body to that of its mother. The breastfeeding duration will be measured with a chronometer in the breastfeedings at these measurement hours. In order to determine the breastfeeding time, after the mother and baby are positioned, the stopwatch will be started when the baby takes the first breast into his mouth. Data collection forms will be filled.
  Interventions: Other: Giving a biological breastfeeding position
- Experimental ( armpit / football breastfeeding position): (Experimental): The first breastfeeding after birth will take place within the first half hour - two hours.The second breastfeeding will be performed 2 hours after the first breastfeeding, and the third breastfeeding will be performed at the 24th hour.Three measurements will be made in total.The baby's head is placed on the breast that is breastfed and the feet are laid flat so that they pass under the armpit of the breastfed side.While the mother's hand on the breastfeeding side holds the baby's head, the other hand directs the breast towards the baby and breastfeeding is initiated.The breastfeeding duration will be measured with a chronometer in the breastfeedings at these measurement hours.In order to determine the breastfeeding time, after the mother and baby are positioned, the stopwatch will be started when the baby takes the first breast into his mouth. Data collection forms will be filled.
  Interventions: Other: Giving a football ( armpit) position

INTERVENTIONS:
Other: Giving a biological breastfeeding position — The mother is half-sitting, in the most comfortable position where she can make eye contact with her baby. The baby's head is placed on the mother's chest with her legs on the mother's stomach. With this position, gravity fixes the baby's whole body to that of its mother.
  Arms: Experimental Group : (Biological Breastfeeding Position)
Other: Giving a football ( armpit) position — The mother sits upright, leaning back, and the baby's bottom and the right or left side of the mother is supported by pillows from whichever side she will breastfeed. The baby's head is placed on the breast that is breastfed and the feet are laid flat so that they pass under the armpit of the breastfed side. While the mother's hand on the breastfeeding side holds the baby's head, the other hand directs the breast towards the baby and breastfeeding is initiated.
  Arms: Experimental ( armpit / football breastfeeding position):

SUMMARY:
Breast milk is a natural, unique, ideal food that best meets the nutritional needs of babies for healthy growth and development. Studies clearly demonstrate the short and long-term benefits of breast milk to the baby, mother, family, environment, economy and country with strong evidence. There are many factors that affect breastfeeding. One of these factors is breastfeeding techniques. Proper breastfeeding technique includes holding the baby well and attaching the baby to the breast correctly, and ineffective breastfeeding techniques, incorrect position and holding style cause poor breastfeeding outcomes in mothers. There are many different breastfeeding positions such as cradle position, cross cradle position, football grip position (armpit position), side-lying breastfeeding, biological breastfeeding. It is of great importance to consider in detail the superiority of these positions over each other. Reveal the advantages of different positions will help increase breastfeeding rates and long-term breastfeeding rates. The aim of this study is to reveal which position is more effective in terms of the effects of biological breastfeeding and armpit (football) breastfeeding positions on breastfeeding self-efficacy, breastfeeding success, breastfeeding duration and postpartum comfort.

The Hypotheses of the Study Hypothesis 0 (H0): There is no difference between biological breastfeeding and armpit (football) breastfeeding position on breastfeeding success, breastfeeding self-efficacy and postpartum comfort in primiparous mothers.

Hypothesis 1 (H1): Breastfeeding success of primiparous mothers in the biological breastfeeding position is higher than in the armpit (football) breastfeeding position.

Hypothesis 2 (H2): Breastfeeding self-efficacy of primiparous mothers in the biological breastfeeding position is higher than in the armpit (football) breastfeeding position.

Hypothesis 3 (H3): Breastfeeding duration of primiparous mothers in the biological breastfeeding position is higher than in the armpit (Football) breastfeeding position.

Hypothesis 4 (H4): Primiparous mothers have higher comfort in the biological breastfeeding position than in the armpit (Football) breastfeeding position.

DETAILED DESCRIPTION:
Breast milk is a natural, unique, ideal food that best meets the nutritional needs of babies for healthy growth and development. Breastfeeding, which has no alternative for the future of societies and the planet, is a fundamental public health priority and goal for all countries. Breast milk is more than just a form of nutrition for the baby. It provides immunity against the vulnerable and immature systems of the newborn and helps protect against many common childhood diseases, both infectious and non-communicable. In addition to protecting children's health, breast milk has the potential to protect women's health and save their lives. Studies clearly demonstrate the short and long-term benefits of breast milk to the baby, mother, family, environment, economy and country with strong evidence .

According to the World Health Organization (WHO), initiating breastfeeding within the first hour is one of the basic neonatal care and should cover every newborn. At the same time, it is recommended to give only breast milk in the first 6 months of life, to continue breastfeeding at 2 years of age and beyond, and to give nutritionally sufficient and safe complementary foods at 6 months. Worldwide, 44% of infants aged 0-6 months were exclusively breastfed in the 2015-2020 period. One of the goals of WHO in its comprehensive implementation plan on maternal, infant and young child nutrition is to increase the rate of exclusive breastfeeding in the first 6 months to at least 50% by 2025. Breastfeeding is not just a physiological event, it is a process that needs to be learned. In this respect, it is of great importance to determine the factors affecting breastfeeding and to deal with successful breastfeeding elements in detail. Successful breastfeeding is a scientifically based art. Proper breastfeeding technique includes holding the baby well and properly attaching the baby to the breast. Ineffective breastfeeding techniques, wrong position and holding style are among the factors that cause poor breastfeeding outcomes in mothers.

There is no standard breastfeeding position, as every mother and baby is special and very different. There are many positions that can be used while breastfeeding. These; cradle, cross cradle, football hold (armpit hold), side-lying breastfeeding, biological breastfeeding positions. There are different studies that compare breastfeeding positions.

It was observed that the mothers in the side lying position were more satisfied with comfort, easy positioning and long-term breastfeeding than the biological nutrition group. In a study comparing reported to pose a low risk three different breastfeeding positions, the football position has been found to be the most biomechanically efficient and has been reported to pose less risk for musculoskeletal disorders in the football position compared to the cradle and cross-cradle positions.In a quasi-experimental study conducted to investigate the effect of biological breastfeeding position on post-cesarean pain, it was observed that moderate post-cesarean pain decreased to mild after biological feeding.

Based on this information, the study was planned to determine the effect of two different breastfeeding positions on breastfeeding success, breastfeeding self-efficacy and postpartum comfort in primiparous mothers.

Method: The population of the study will be composed of primiparous mothers who gave birth in Bursa City Hospital and who were hospitalized in the Gynecology and Obstetrics Clinics between July 2023 and November 2024. The sample will consist of mothers who voluntarily accepted to participate in the study and who met the inclusion criteria of the study between the specified dates. The effect width value was taken as 0.70 as the method used when it was not known how many units difference between the groups was significant. The effect width value gives results of with 0.20 a very high constraint, 0.50 at medium level, and 0.80 under the maximum acceptance constraint. In the case where the 5% tolarance and the 80.15% power level, the effect width value is 0.70, the total number of mothers-infants was determined as 68, including 34 control and 34 experimental groups, which met the inclusion criteria of the research.

Pregnant women will be informed about the purpose of the study, how to collect, store and use data. Verbal and written consents will be obtained from the pregnant women who accept to participate in the study by filling in the "Informed Voluntary Consent Form". Pre-breastfeeding Mother Descriptive Information Form, Newborn Descriptive Information Form, Postpartum Breastfeeding Self-Efficacy Short Form, Postpartum Comfort Scale will be filled face to face with the mother. The first breastfeeding after birth will take place within the first half hour - two hours. The second breastfeeding will be performed 2 hours after the first breastfeeding, and the third breastfeeding will be performed at the 24th hour. Three measurements will be made in total. The breastfeeding duration will be measured with a chronometer in the breastfeedings at these measurement hours. In order to determine the breastfeeding time, after the mother and baby are positioned, the stopwatch will be started when the baby takes the first breast into his mouth. Breastfeeding Scoring System (LATCH) and Postpartum Comfort Scale will be filled in by supporting and observing breastfeeding at each measurement. The LATCH scale will be completed by two observers during breastfeeding. In the last measurement, the Breastfeeding Self-Efficacy Scale will also be filled in. After breastfeeding, the baby's gas will be removed and it will be supported to be in a comfortable and safe position and the mother will be rested.

ELIGIBILITY:
Inclusion Criteria:

Mother's Inclusion Criteria:

* Be over the age of 19
* Able to speak Turkish language
* Without any communication problems and collaborative
* Absence of any complications in pregnancy such as multiple pregnancy, preeclampsia, gestational diabetes, ablation placenta.
* Having a normal vaginal birth
* Having a term and primiparous (singular) baby
* Breast milk is not contraindicated to the baby
* Absence of nipple problems that will affect breastfeeding
* No previous breastfeeding experience Newborn's Inclusion Criteria
* Such as craniofacial anomaly such as cleft palate, cleft lip, paralysis of facial muscles, etc. absence of congenital anomalies that would prevent sucking
* APGAR score of 7 or higher in the 5th minute
* Having "sucking, swallowing and breathing coordination"

Exclusion Criteria:

Mother's Exclusion Criteria:

* Refusal to participate in the study
* Not signing the informed consent form
* Having a communication problem
* Desire to leave at any stage of the study or early discharge
* Postpartum bleeding, infection, etc. development in the mother
* Not being able to take the desired position for some reason, having a physical disability

Newborn's Exclusion Criteria:

* Transfer to another centre
* Developing a complication such as respiratory distress

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 68 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
The effect of Group 1 (biological breastfeeding position) and Group 2 (armpit / football breastfeeding position) on breastfeeding self-efficacy. | Within postpartum 24th hour
  (Breast-Feeding Self-Efficacy Scale- Short Form/BSES-SF): (Breast-Feeding Self-Efficacy Scale- Short Form/BSES-SF): Breastfeeding Self-Efficacy Scale is a 33-item scale developed by Dennis and Faux in 1999. The Breastfeeding Self-Efficacy Scale Short Form was developed by Dennis (2003) by reducing it to a 14-item scale. The validity and reliability of the scale in our country was done by Tokat Aluş, Okumus, and Dennis (2010). The scale is a 5-point Likert-type scale and is evaluated as I am never sure (1 point) and I am always sure (5 points). The minimum score that can be obtained from the scale is 14, and the maximum score is 70. The scale has no breakpoints. An increase in the scale score means higher breastfeeding self-efficacy. The cronbach alpha value of the scale was found to be 0.87.
The effect of Group 1 (biological breastfeeding position) and Group 2 (armpit / football breastfeeding position) on breastfeeding success. | Within postpartum 24th hour
  LATCH : Jensen et al. (1994) provides a systematic evaluation of breastfeeding and the identification of areas that require intervention in breastfeeding. Each letter of the abbreviation LATCH indicates a breastfeeding assessment area.
  * "L" baby's ability to grasp the breast,
  * "A" The presence of baby audible swallowing at the breast,
  * "T" mother's nipple type,
  * "C" is the mother's sense of comfort,
  * "H" refers to the position the mother uses to hold or breastfeed, and the amount of help the mother needs to hold the baby.
  Scale evaluation is done by giving 0, 1 and 2 points to each item. Breastfeeding success is evaluated by summing the scores. The highest score that can be obtained from the scale is 10 and the lowest score is 0. An increase in the scores obtained from the scale indicates the success of breastfeeding.

SECONDARY OUTCOMES:
The effect of Group 1 (biological breastfeeding position) and Group 2 (armpit / football breastfeeding position) on postpartum comfort. | Within postpartum 24th hour
  Postpartum Comfort Scale: The postpartum comfort scale was developed by Karakaplan and Yıldız in 2010. It was developed to evaluate the postpartum comfort of mothers who had cesarean section or normal vaginal delivery in a holistic approach based on the comfort theory and is used to evaluate the physical, psychospiritual, sociocultural and environmental comforts of mothers as a whole.The scale consists of 34 items.. The average value is determined by dividing the total score obtained from the scale by the number of items, and the result is shown in the 1-5 distribution. Basically, low comfort is expressed with 1 and high comfort with 5. The lowest score to be taken from the scale is 34 and the highest score is 170. An increase in the total score obtained from the scale indicates that the comfort level is high.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Menekşe, Asist.Prof., Study Director — Sakarya University; Sema Aktaş, Nurse, Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiryaki Ö., Pekşen S. (2019). Anne Sütü ve Emzirme; Anneler Sordu Biz Cevapladık. Editör: Çınar N. Ankara:Gece Akademi. s. 26-30
- [Background] Doherty T, Horwood C, Pereira-Kotze C, du Plessis L, Witten C. Stemming commercial milk formula marketing: now is the time for radical transformation to build resilience for breastfeeding. Lancet. 2023 Feb 11;401(10375):415-418. doi: 10.1016/S0140-6736(23)00095-8. Epub 2023 Feb 7. No abstract available. PMID 36764312
- [Background] Christian P, Smith ER, Lee SE, Vargas AJ, Bremer AA, Raiten DJ. The need to study human milk as a biological system. Am J Clin Nutr. 2021 May 8;113(5):1063-1072. doi: 10.1093/ajcn/nqab075. PMID 33831952
- [Background] Duan X, Wang J, Jiang X. A meta-analysis of breastfeeding and osteoporotic fracture risk in the females. Osteoporos Int. 2017 Feb;28(2):495-503. doi: 10.1007/s00198-016-3753-x. Epub 2016 Aug 30. PMID 27577724
- [Background] WHO. (2020). Newborns: improving survival and well-being. https://www.who.int/news-room/fact-sheets/detail/newborns-reducing-mortality Erişim Tarihi: 05.03.2023
- [Background] WHO, (2021). Infant and young child feding. https://www.who.int/news-room/fact-sheets/detail/infant-and-young-child-feeding Erişim Tarihi: 05.03.2023
- [Background] Çınar N., Şahin S. (2020) Anne ve Çocuk Sağlığı ilk 1000 gün. Akademisyen Kitabevi. Ankara. S:264
- [Background] Colson S. 2018. Biological nurturing; İnstinctual Breastfeeding. Foreword by Kerstin Uvnas Moberg; 2 nd revised and uodated edition, London, Pinter & Martin, 4-148.
- [Background] Davra, K., Chavda, P., Pandya, C., Dave, D., & Mehta, K. (2022). Breastfeeding position and attachment practices among lactating mothers: An urban community-based cross-sectional study from Vadodara city in western India. Clinical Epidemiology and Global Health, 15, 101009.
- [Background] Colson SD, Meek JH, Hawdon JM. Optimal positions for the release of primitive neonatal reflexes stimulating breastfeeding. Early Hum Dev. 2008 Jul;84(7):441-9. doi: 10.1016/j.earlhumdev.2007.12.003. Epub 2008 Feb 19. PMID 18243594
- [Background] WHO. (2023). Erişim adresi: https://www.who.int/health-topics/breastfeeding#tab=tab_1 Erişimtarihi: 05.03.2023.
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Ezeukwu OA, Ojukwu CP, Okemuo AJ, Anih CF, Ikele IT, Chukwu SC. Biomechanical analysis of the three recommended breastfeeding positions. Work. 2020;66(1):183-191. doi: 10.3233/WOR-203162. PMID 32417825
- [Background] Reni, C., Sinar, P., & Etin, R. (2020). Effect of Biologic Nurturing Baby Led Feeding on Post Sectio Caesarea Pain Scale In Majenang Hospital 2018. Midwifery And Nursing Research (MANR) Journal, 2(1), 22-27.
- [Background] Puapornpong P, Raungrongmorakot K, Laosooksathit W, Hanprasertpong T, Ketsuwan S. Comparison of Breastfeeding Outcomes Between Using the Laid-Back and Side-Lying Breastfeeding Positions in Mothers Delivering by Cesarean Section: A Randomized Controlled Trial. Breastfeed Med. 2017 May;12:233-237. doi: 10.1089/bfm.2016.0193. Epub 2017 Apr 6. PMID 28384091